CLINICAL TRIAL: NCT04690842
Title: Implementation of PTH Measurement Intra / Post Thyroidectomy to Improve Post Surgical Safety in Pediatric Patients
Brief Title: Improving Safety in Pediatric Thyroidectomy by PTH Measurements
Status: Completed | Type: Observational
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Analía Freire, Pediatric Endocrinology, PhD, Hospital de Niños R. Gutierrez de Buenos Aires
Other Study IDs: CEI 19.27
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Hypoparathyroidism Postprocedural
Keywords: Thyroidectomy; PTH; Pediatric surgery; hypocalcemia
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PTH measurements post-thyroidectomy (at 5 and 60 min post thyroid removal) — We implement an algorithm employing PTH levels post-thyroidectomy to stratify patients according to their postsurgical risk for hypoparathyroidism, and to distinctively manage them in the immediate postsurgical period. High risk patients are quickly supplemented with Calcium iv and activated 25OH vitamin D. Low risk patients are clinically controlled and calcium level were checked at 24 and 48 hs post thyroidectomy.

SUMMARY:
We implemented a previously reported algorithm based on intra-postoperative PTH measurements with selected cut-off values, both to predict post-thyroidectomy hypoparathyroid hypocalcemia, and to guide postsurgical management. The objective of the study was to assess if this strategy was useful to reduce hypocalcemia, post-surgery calcium sampling and hospitalization length.

DETAILED DESCRIPTION:
Sixty-six patients were included in the analysis. Based on their intra-operatory PTH determinations, patients were classified according to their post-surgical hypoparathyroidism risk and were either immediately treated with calcium and vitamin D1-25 supplementation (high-risk) or assigned to clinical control and routine calcium sampling (low-risk). The outcomes and overall results of these therapeutical approaches were compared with those of a control group, started on treatment when TCa levels dropped below normal.

In the high-risk subgroup (n=30) five patients showed hypocalcemia within the first 24 hours. Compared with the high-risk control subgroup, the incidence of hypocalcemia fell from 100% to 17% (p<0.001), and the median hospitalization length from 6 to 3 days (p<0.001).

In the low-risk subgroup (n=36) 28 patients remained normocalcemic with significantly less calcium sampling (p<0.001). Eight patients had hypocalcemia; 7 of them required neck dissection, which was the only risk factor related to post-surgical hypoparathyroidism (RR: 2.1 [CI 95% 1.4-3.1], P<0.001).

Compared to the control group, overall incidence of hypocalcemia was reduced by 58 %.

This approach improved patient's safety by reducing the occurrence of hypocalcemia and the length of hospitalization after thyroidectomy in pediatric patients. Preventive calcium supplementation seems to be more beneficial in patients undergoing neck dissection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent total thyroidectomy between January 2014 and April 2020

Exclusion Criteria:

* Patients with known hyper or hypoparathyroidism, kidney failure, and those taking medications known to affect TCa, PTH, or vitamin D levels (octreotide, oral glucocorticoids, diuretics and antiepileptics), or any other condition that could interfere with calcium metabolism

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients between 2 and 19 years of age who underwent total thyroidectomy at Hospital de Niños Ricardo Gutiérrez in Buenos Aires, Argentina between January 2014 and April 2020 were included. Exclusion criteria were patients with known hyper or hypoparathyroidism, kidney failure, and those taking medications known to affect TCa, PTH, or vitamin D levels (octreotide, oral glucocorticoids, diuretics and antiepileptics), or any other condition that could interfere with calcium metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Biochemical hypocalcemia post thyroidectomy occurrence | 48 hours postthyroidectomy
  total Calcium level < 8 mg/dl
Symptomatic hypocalcemia post thyroidectomy ocurrence | 48 hours posthyroidectomy
  Signs o symptoms of hypocalcemia (Chvostek or Trousseau signs, tingling, numbness, muscle cramps, spasms, tetany or seizures

SECONDARY OUTCOMES:
days of hospitalization after thyroidectomy | up to 15 days after thyroidectomy
  number of days that patient need hospitalization (high risk group)
number of Calcium sampling | 48 hours postthyroidectomy
  number of venipuncture performed to control serum calcium level (low risk group)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freire AV, Ropelato MG, Ballerini MG, Acha O, Bergada I, de Papendieck LG, Chiesa A. Predicting hypocalcemia after thyroidectomy in children. Surgery. 2014 Jul;156(1):130-6. doi: 10.1016/j.surg.2014.02.016. Epub 2014 Feb 27. PMID 24929763